CLINICAL TRIAL: NCT06040151
Title: Evaluating Mobile-based Medication Reconciliation by Patients at Home: Feasibility, Quality and Time Investments by Pharmacy Technicians
Brief Title: Evaluating Mobile-based Medication Reconciliation by Patients at Home
Acronym: PILLS@HOME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Alan Abdulla, dr. Alan Abdulla, Principal Investigator, Erasmus Medical Center
Other Study IDs: 10624
Record Dates: First submitted 2023-07-12; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Patients
Keywords: Patients with all conditions are eligible

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users of mobile-based medication-reconciliation app: Adult patients (18 years or older) who are asked to complete medication reconciliation before a planned admission to the clinical ward of selected pilot departments in Erasmus Medical Center
  Interventions: Device: Digizorg mobile app (quality evaluation study)

INTERVENTIONS:
Device: Digizorg mobile app (quality evaluation study) — Erasmus Medical Center is developing a state-of-the-art, mobile-based patient portal that combines up-to-date medication lists from all healthcare providers involved in a patient's care. Other functionalities include: accessing health information, viewing and planning appointments, teleconsulting, sending messages, filling in questionnaires, reporting self-measurements, and reading background information on diseases, medication, and other interventions. The patient portal will primarily be implemented in Erasmus Medical Center, and is ultimately intended for every patient, regardless of underlying condition.

SUMMARY:
Medication reconciliation (MR) is essential to limit drug-related problems that occur during care transitions in and out of care institutions. Pharmacy-led medication reconciliation has been shown to reduce medication discrepancies, preventable harm and hospital readmissions. However, these consultations are time-consuming. The Erasmus Medical Center is currently developing a mobile-based patient portal. After receiving an invitation to perform medication reconciliation in the app, patients can review their medication and allergies at home. Next, pharmacy technicians manually verify all patient-entered data on completeness and quality. The investigators hypothesize that mobile-based medication reconciliation results in increased patient insight. Yet, it is unknown if mobile-based medication reconciliation is feasible, saves time, and is of high quality.

Therefore, the primary study objectives are to assess (1) the feasibility of patients performing medication reconciliation using a mobile-based patient portal, (2) the time investment of pharmacy technicians in mobile-based medication reconciliation (and related costs), in comparison to standard practice, and (3) the quality of patients' pre-verified medication lists. The secondary study objective is to assess patients' and pharmacy technicians' acceptability of performing medication reconciliation using a mobile-based patient portal.

This is a prospective quality evaluation study assessing mobile-based medication reconciliation. All adult patients (18 years or older) who are admitted to (a selection of) clinical ward in Erasmus Medical Center and who are asked to complete medication reconciliation are eligible. In the patient app, patients review ('pre-verify') their medications and allergies, after which pharmacy technicians check and manually approve ('verify') all patient-entered data and determine whether a follow-up interview is needed.

Feasibility is defined as the successful completion rate of digital medication reconciliation, and the need for additional interviews. Time investment by pharmacy technicians (and related costs) are determined by timing the duration of all patient-bound medication reconciliation-related tasks, both in standard care and when using mobile-based reconciliation. The quality of verification is determined by comparing patients' pre-verified medication list to pharmacy technician-verified lists. Acceptability is defined as the perceived usability of medication reconciliation by patients and by pharmacy technicians.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Planned admission to the clinical ward of participating pilot departments in Erasmus MC

Exclusion Criteria:

* No potential subject will be excluded from participation in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients (18 years or older) who are asked to complete medication reconciliation before a planned admission to the clinical ward of selected pilot departments in Erasmus MC are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility (1/4): completion rate of digital MR by patients | During quality evaluation of the patient app, an average of 3 months
  The fraction of all patients who were invited to participate that participated
Feasibility (2/4): the time it takes patients to perform digital MR (in minutes) | During quality evaluation of the patient app, an average of 3 months
  To assess the ease-of-use of performing medication reconciliation in the patient app
Feasibility (3/4): the need for live, follow-up interviews after performing digital MR | During quality evaluation of the patient app, an average of 3 months
  The fraction of all patients who were invited to participate in digital MR who needed a live interview
Feasibility (4/4): how often the helpdesk was contacted | During quality evaluation of the patient app, an average of 3 months
  The fraction of all patients who were invited to participate in digital MR who contact the helpdesk
The time investment by pharmacy technicians per patient in the digital MR process, compared to the current situation (in minutes) | Before launch of the patient app, during an average of 2 months, and during quality evaluation of the patient app, an average of 3 months
  The time investment by pharmacy technicians per patient in the new workflow vs. the current situation, in which all patients are invited for a live interview
The quality of a patient's pre-verified medication list, compared to the pharmacy technician's verified medication list | During quality evaluation of the mobile-based medication reconciliation tool, an average of 3 months
  The number of discrepancies between the patient-reported medication list and the pharmacy-verified medication list (the number of changes made by a pharmacy technician in the MR process)

SECONDARY OUTCOMES:
Acceptability (1/2): defined as the perceived usability of mobile-based MR by patients, assessed using short in-app questionnaires (VAS 1-5) | During quality evaluation of the mobile-based medication reconciliation tool, an average of 3 months
  To assess to what extent digital medication reconciliation is accepted by patients
Acceptability (2/2): defined as the perceived usability of mobile-based MR by patients and pharmacy technicians, assessed using short qualitative interviews with both patients and pharmacy technicians | During quality evaluation of the mobile-based medication reconciliation tool, an average of 3 months
  To assess to what extent digital medication reconciliation is accepted by patients and pharmacy technicians

IPD SHARING:
Plan to Share IPD: Undecided